CLINICAL TRIAL: NCT04737629
Title: Understanding the Effects of Herbs on Attention, Coordination, and Taste
Brief Title: Understanding the Effects of Water-related Appetite Expectancies on Caloric Intake in College Students
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never started.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB202001347
Record Dates: First submitted 2021-01-21; First posted 2021-02-04 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Appetitive Behavior; Weight Loss; Water; Energy Intake
MeSH Terms: conditions — Appetitive Behavior; Weight Loss | interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Expectancy and Water Condition (Experimental)
  Interventions: Behavioral: Expectancy and Water
- No Expectancy and Water Condition (Experimental)
  Interventions: Behavioral: No Expectancy and Water
- No Water Condition (Experimental)
  Interventions: Behavioral: No Water

INTERVENTIONS:
Behavioral: Expectancy and Water — In the expectancy and water condition, participants will be instructed to consume the mint herb and 500mL of water before the start of the taste test. The script for this condition will inform them of research that has shown water to decrease appetite by up to 50% (attempting to create an expectancy).
  Arms: Expectancy and Water Condition
Behavioral: No Expectancy and Water — Participants will be instructed to consume the mint herb and 500mL of water before the start of the taste test. The script will inform them of research that has shown water to decrease appetite by up to 50%. In this condition, however, the research team will also inform them that this herb is expected to counteract the effects of water on appetite because it decreases water retention, causing water to pass through the stomach and intestines at a faster than normal rate (attempting to create no water expectancy or nullify any pre-existing expectancy).
  Arms: No Expectancy and Water Condition
Behavioral: No Water — Participants will be instructed to consume the mint herb and 50mL of water before the start of the taste test. Participants will be given 100mL of water during the taste test to aid in their ability to taste and consume food, and to avoid acute thirst interfering with food consumption. Access to fluids during a taste test has been used in control conditions in similar studies. The script for this condition will inform participants of research that has shown water to decrease appetite by up to 50% but acknowledge that they will not be receiving water (thus, they should not expect an effect on appetite).
  Arms: No Water Condition

SUMMARY:
Consuming large volumes of water has recently been identified as a common weight loss strategy among U.S. adults. It is a widespread belief that drinking water increases feelings of satiety and reduces food intake, which could contribute to long-term weight maintenance. Many studies have shown support for this, demonstrating water's ability to reduce hunger and energy intake. In some cases, increased water consumption was associated with weight loss. However, the mechanisms of how water affects food intake have been minimally explored. There is potential that the effect of water on reduced food intake and increased satiety is due to individuals' belief that water will reduce their appetite and food intake. The question remains if water expectancy has a meaningful influence on water's ability to reduce food intake. The investigators hypothesize that participants will report less hunger and consume fewer calories when given water and an expectancy that water will affect appetite, compared to a condition when given water and do not expect water to have an effect on appetite. We further hypothesize that calorie intake will not meaningfully differ when participants are given water with no expectancies compared to when given no water. During this experiment, the investigators will vary the presence of water and manipulate expectancies about water's effects on appetite across three conditions: (1) an expectancy and water condition; (2) an expectancy and no water condition; and (3) a no expectancy and water condition. In each condition, participants will engage in a bogus taste test and complete two short cognitive tasks for distraction purposes. In an effort to prevent demand characteristics, this study involves deception. Participants will be told that the research team is interested in testing the effects of three different mint herb variations on attention, coordination, and taste perceptions. After completing the cognitive tasks and taste test, participants will have a 10 minute period to eat as much of the remaining food as they'd like. Food will be weighed before and after this period (without the participant's knowledge) in order to determine caloric intake.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years of age
* rating at least two foods from each category (chips/crackers and sweets/candies) on the food options list for the taste test as a 7 ("like moderately") or higher on a 9-point hedonic scale
* willing/able to come to the lab for three sessions

Exclusion Criteria:

* current smoker
* self-report of a current or past eating disorder diagnosis
* taking an appetite suppressant or stimulant medication
* currently engaged in a weight loss program
* currently pregnant, breastfeeding, or planning to become pregnant
* allergy to mint

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Caloric intake | Through study completion, up to 9 weeks.
  Weighing food on digital food scale after taste test.

SECONDARY OUTCOMES:
Appetite | Through study completion, up to 9 weeks.
  Four-question 100mm visual analog scale (VAS) assessing assesses hunger, fullness, satiety, and prospective food consumption. The minimum possible score is 0, and the maximum possible score is 100.
Physical activity | Assessed at baseline before any experiment administration.
  International Physical Activity Questionnaire (IPAQ-SF). Participants are categorized into low, moderate, or high levels of physical activity. Higher score indicates more physical activity engagement (better outcome).
Restrained eating | Assessed at baseline before any experiment administration.
  Eating Disorder Examination Questionnaire (EDE-Q). The minimum possible score is 0 and maximum possible score is 34.5. A higher score indicates higher restrained eating symptoms (poorer outcome).
Habitual water intake | Assessed at baseline before any experiment administration.
  As part of the baseline questionnaire, participants will be asked about how many glasses of water they drank over the past 7 days in order to assess habitual water intake. Response options range from "I did not drink water during the past 7 days" to "4 or more glasses per day."

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared on the Open Science Framework (OSF) platform following the completion of the study. The study protocol, statistical analysis plan, and de-identified analytic code will be available.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available within 12 months following the completion of the study.
Access Criteria: No access criteria. De-identified data will be available to anyone.

REFERENCES:
- [Background] Han L, You D, Zeng F, Feng X, Astell-Burt T, Duan S, Qi L. Trends in Self-perceived Weight Status, Weight Loss Attempts, and Weight Loss Strategies Among Adults in the United States, 1999-2016. JAMA Netw Open. 2019 Nov 1;2(11):e1915219. doi: 10.1001/jamanetworkopen.2019.15219. PMID 31722029
- [Background] Lappalainen R, Mennen L, van Weert L, Mykkanen H. Drinking water with a meal: a simple method of coping with feelings of hunger, satiety and desire to eat. Eur J Clin Nutr. 1993 Nov;47(11):815-9. PMID 8287852
- [Background] Davy BM, Dennis EA, Dengo AL, Wilson KL, Davy KP. Water consumption reduces energy intake at a breakfast meal in obese older adults. J Am Diet Assoc. 2008 Jul;108(7):1236-9. doi: 10.1016/j.jada.2008.04.013. PMID 18589036
- [Background] Daniels MC, Popkin BM. Impact of water intake on energy intake and weight status: a systematic review. Nutr Rev. 2010 Sep;68(9):505-21. doi: 10.1111/j.1753-4887.2010.00311.x. PMID 20796216
- [Background] Dennis EA, Dengo AL, Comber DL, Flack KD, Savla J, Davy KP, Davy BM. Water consumption increases weight loss during a hypocaloric diet intervention in middle-aged and older adults. Obesity (Silver Spring). 2010 Feb;18(2):300-7. doi: 10.1038/oby.2009.235. Epub 2009 Aug 6. PMID 19661958
- [Background] Corney RA, Sunderland C, James LJ. Immediate pre-meal water ingestion decreases voluntary food intake in lean young males. Eur J Nutr. 2016 Mar;55(2):815-819. doi: 10.1007/s00394-015-0903-4. Epub 2015 Apr 18. PMID 25893719
- [Background] Stookey JJ. Negative, Null and Beneficial Effects of Drinking Water on Energy Intake, Energy Expenditure, Fat Oxidation and Weight Change in Randomized Trials: A Qualitative Review. Nutrients. 2016 Jan 2;8(1):19. doi: 10.3390/nu8010019. PMID 26729162
- [Background] Madjd A, Taylor MA, Delavari A, Malekzadeh R, Macdonald IA, Farshchi HR. Effects on weight loss in adults of replacing diet beverages with water during a hypoenergetic diet: a randomized, 24-wk clinical trial. Am J Clin Nutr. 2015 Dec;102(6):1305-12. doi: 10.3945/ajcn.115.109397. Epub 2015 Nov 4. PMID 26537940
- [Background] Casazza K, Brown A, Astrup A, Bertz F, Baum C, Brown MB, Dawson J, Durant N, Dutton G, Fields DA, Fontaine KR, Heymsfield S, Levitsky D, Mehta T, Menachemi N, Newby PK, Pate R, Raynor H, Rolls BJ, Sen B, Smith DL Jr, Thomas D, Wansink B, Allison DB. Weighing the Evidence of Common Beliefs in Obesity Research. Crit Rev Food Sci Nutr. 2015;55(14):2014-53. doi: 10.1080/10408398.2014.922044. PMID 24950157